CLINICAL TRIAL: NCT06501508
Title: Abdominal Wall Dehiscence After Laparotomy Closure in Abdominal Surgery: a Retrospective Observational Study on the Influence of the Suture Used
Acronym: SUTURA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PIC089-23_FJD
Record Dates: First submitted 2023-11-22; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-11

CONDITIONS: Surgical Wound Dehiscence
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Stratafix: All patients in which Stratafix symmetric was used for the primary closure of the abdominal wall incision
  Interventions: Device: Stratafix Symmetric
- Control: All patients in which other, conventional suture types were used for primary closure of the abdominal wall incision

INTERVENTIONS:
Device: Stratafix Symmetric — Use of Stratafix Symmetric for primary fascial closure
  Groups: Stratafix

SUMMARY:
In this retrospective longitudinal observational study we compare the incidence of fascial dehiscence and incisional hernia in patients operated via abdominal wall incision, comparing the barbed suture Stratafix Symmetric to other types of suture during closure of the abdominal wall. In addition, we plan to analize the impact of other risk factors, patient related and patient unrelated, on the incidence of fascial dehiscence.

DETAILED DESCRIPTION:
In this retrospective longitudinal observational study we primarily aim to compare the influence of the applied suture type (Stratafix Symmetric versus other suture types) for primary fascial closure in abdominal surgery on the incidence of fascial dehiscence.

Secondary outcomes such as will also be analized. Primary outcomeis the incidence of abdominal wall dehiscence. Secondary outcomes are the impact of the occurrence of abdominal wall dehiscence on mortality and hospital stay, the influence of other risk factors on the occurrence of abdominal wall dehiscence, the influence of the suture type and other risk factors on the incidence of incisional hernia after 12 months of follow-up and a speciality subgroup analysis.

The diagnoses of each patient and the procedures performed are coded according to ICD 9 or ICD 10. For primary cause diagnoses and secondary diagnoses, external causes and procedures, ICD9/ICD10 codes are also used. Following the AHQR definition, cases of laparotomy dehiscence will be defined as those whose ICD 9/ICD 10 codes conform to "New closure of postoperative abdominal wall disruption", as well as those identified secondarily after crossing the databases as reoperated for this reason with another coding.

Statistical analysis will be performed using statistical techniques appropriate to the variables under study. A descriptive analysis of the population will be performed, frequency results will be expressed in absolute terms, such as percentages and confidence intervals. The percentage of subjects with dehiscence will be calculated by the group. A two-sided 95% confidence interval (CI) for the difference in percentages (Stratafix - Control) will be estimated using the Wald method. If the upper limit of the confidence interval for the difference in percentages (Stratafix-Control) is below 0, then it will be concluded that the true dehiscence rate for Stratafix is lower than that for the control. In addition, two-sided 95% CIs within each group will be estimated for the dehiscence rate using the Clopper-Pearson method.

Continuous variables will be expressed as mean (SD) and median (range) according to the normality test (Kolmogorov Smirnov test). For the study of the relationship between the different variables, Chi-square or Analysis of Variance will be used if they are parametric. And if they do not follow a normal distribution, nonparametric tests will be used (Mann-Whitney U or Kruskal Wallis, as appropriate). Biochemical recurrence-free survival (BCR-free survival) will be estimated using Kaplan-Meier curves. SPSS. 21 (SPSS Inc. Chicago, IL, USA) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years, abdominal incision or laparoscopy with extraction site incision

Exclusion Criteria:

* Pregnancy, use of mesh for fascial closure in primary surgery, history of ventral abdominal hernia surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults over 18 years of age operated via laparotomy or laparoscopy with extraction site incision in the 4 participating Hospitals between 01/01/2018 and 21/11/23
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2024-11-22 (Estimated)

PRIMARY OUTCOMES:
Abdominal Wall Dehiscence | 30 days
  Disruption of all layers of the abdominal wall with exposure of abdominal viscera within 30 days after primary surgery

SECONDARY OUTCOMES:
Incisional hernia | 1 year
  Any defect of the abdominal wall in the area of the primary incision, palpable or visible in ultrasound, CT- or MR-Scan, with or without protrusion of intraabdominal content
PROMs - Postoperative Pain | 1 year
  One question about pain - 4 answers
PROMs - Mental and emotional health | 1 year
  Two questions - 4 answers for each question
PROMs - Work an social life performance | 1 year
  Two questions - 4 answers for each question
PROMs - Fatigue | 1 year
  Two questions - 4 answers for each question
PROMs - Funcionality | 1 year
  One question - 4 answers for each question
PROMs - Sexuality | 1 year
  One question - 4 answers for each question
PROMs - Body image | 1 year
  One question - 4 answers for each question

CONTACTS AND LOCATIONS:
Overall Officials: Hector Gauadalajara Labajo, PHD, Principal Investigator — Quironsalud
Locations (4):
- Spain (4):
  - Hospital universitario General de Villalba, Collado Villalba, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zolin SJ, Rosen MJ. Failure of Abdominal Wall Closure: Prevention and Management. Surg Clin North Am. 2021 Oct;101(5):875-888. doi: 10.1016/j.suc.2021.07.001. PMID 34537149
- [Background] Rodriguez-Hermosa JI, Codina-Cazador A, Ruiz B, Roig J, Girones J, Pujadas M, Pont J, Aldeguer X, Acero D. [Risk factors for acute abdominal wall dehiscence after laparotomy in adults]. Cir Esp. 2005 May;77(5):280-6. doi: 10.1016/s0009-739x(05)70854-x. Spanish. PMID 16420934
- [Background] Gili-Ortiz E, Gonzalez-Guerrero R, Bejar-Prado L, Ramirez-Ramirez G, Lopez-Mendez J. [Postoperative dehiscence of the abdominal wound and its impact on excess mortality, hospital stay and costs]. Cir Esp. 2015 Aug-Sep;93(7):444-9. doi: 10.1016/j.ciresp.2015.02.005. Epub 2015 May 6. Spanish. PMID 25956459
- [Background] Jensen KK, Oma E, van Ramshorst GH, Nordholm-Carstensen A, Krarup PM. Abdominal wound dehiscence is dangerous: a nationwide study of 14,169 patients undergoing elective open resection for colonic cancer. Hernia. 2022 Feb;26(1):75-86. doi: 10.1007/s10029-020-02350-z. Epub 2021 Jan 4. PMID 33394254
- [Background] Farquhar M. AHRQ Quality Indicators. In: Hughes RG, editor. Patient Safety and Quality: An Evidence-Based Handbook for Nurses. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Apr. Chapter 45. Available from http://www.ncbi.nlm.nih.gov/books/NBK2664/ PMID 21328764
- [Background] Zucker BE, Simillis C, Tekkis P, Kontovounisios C. Suture choice to reduce occurrence of surgical site infection, hernia, wound dehiscence and sinus/fistula: a network meta-analysis. Ann R Coll Surg Engl. 2019 Mar;101(3):150-161. doi: 10.1308/rcsann.2018.0170. Epub 2018 Oct 5. PMID 30286645
- [Background] Jenkins TP. The burst abdominal wound: a mechanical approach. Br J Surg. 1976 Nov;63(11):873-6. doi: 10.1002/bjs.1800631110. PMID 137024
- [Background] Henriksen NA, Deerenberg EB, Venclauskas L, Fortelny RH, Miserez M, Muysoms FE. Meta-analysis on Materials and Techniques for Laparotomy Closure: The MATCH Review. World J Surg. 2018 Jun;42(6):1666-1678. doi: 10.1007/s00268-017-4393-9. PMID 29322212
- [Background] Patel SV, Paskar DD, Nelson RL, Vedula SS, Steele SR. Closure methods for laparotomy incisions for preventing incisional hernias and other wound complications. Cochrane Database Syst Rev. 2017 Nov 3;11(11):CD005661. doi: 10.1002/14651858.CD005661.pub2. PMID 29099149
- [Background] Cengiz Y, Blomquist P, Israelsson LA. Small tissue bites and wound strength: an experimental study. Arch Surg. 2001 Mar;136(3):272-5. doi: 10.1001/archsurg.136.3.272. PMID 11231844
- [Background] Fortelny RH. Abdominal Wall Closure in Elective Midline Laparotomy: The Current Recommendations. Front Surg. 2018 May 23;5:34. doi: 10.3389/fsurg.2018.00034. eCollection 2018. PMID 29876355
- [Background] Muysoms FE, Antoniou SA, Bury K, Campanelli G, Conze J, Cuccurullo D, de Beaux AC, Deerenberg EB, East B, Fortelny RH, Gillion JF, Henriksen NA, Israelsson L, Jairam A, Janes A, Jeekel J, Lopez-Cano M, Miserez M, Morales-Conde S, Sanders DL, Simons MP, Smietanski M, Venclauskas L, Berrevoet F; European Hernia Society. European Hernia Society guidelines on the closure of abdominal wall incisions. Hernia. 2015 Feb;19(1):1-24. doi: 10.1007/s10029-014-1342-5. Epub 2015 Jan 25. PMID 25618025
- [Background] Tolstrup MB, Watt SK, Gogenur I. Reduced Rate of Dehiscence After Implementation of a Standardized Fascial Closure Technique in Patients Undergoing Emergency Laparotomy. Ann Surg. 2017 Apr;265(4):821-826. doi: 10.1097/SLA.0000000000001762. PMID 28267697
- [Background] Denys A, Monbailliu T, Allaeys M, Berrevoet F, van Ramshorst GH. Management of abdominal wound dehiscence: update of the literature and meta-analysis. Hernia. 2021 Apr;25(2):449-462. doi: 10.1007/s10029-020-02294-4. Epub 2020 Sep 8. PMID 32897452
- [Background] Pereira Rodriguez JA, Amador-Gil S, Bravo-Salva A, Montcusi-Ventura B, Sancho-Insenser JJ, Pera-Roman M, Lopez-Cano M. Small bites technique for midline laparotomy closure: From theory to practice: Still a long way to go. Surgery. 2021 Jul;170(1):140-145. doi: 10.1016/j.surg.2020.12.007. Epub 2021 Jan 15. PMID 33455821